CLINICAL TRIAL: NCT04174287
Title: Modeling the Relationships Between Functional Connectivity and Amyloid Deposition in Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801833A0
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer's Disease
Keywords: 18F-FDG PET scan; amyloid PET; Amyloid beta; Alzheimer's disease; metabolic connectivity; functional connectivity
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — florbetapir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F-18-AV45 (Experimental): F-18-AV45 imaging
  Interventions: Drug: F-18-AV45

INTERVENTIONS:
Drug: F-18-AV45 — The study will enroll 200 patients with prodromal AD and mild AD dementia and 100 normal controls, men and women aged 55-80 years across core clinical criteria of prodromal AD and mild AD dementia based on IWG-2 criteria.

SUMMARY:
Glucose is the main energy source of brain. Different neural degenerative diseases such as Parkinson's disease or Alzheimer's disease have shown distinct brain glucose metabolic patterns. FDG-PET is a established non-invasive method to measures cerebral glucose metabolism and can be used to differentiate different types of neurodegenerative diseases that anatomical imaging such as CT or MRI may not be able to differentiate. Among patients whose Alzheimer's diseases have not been confirmed, the defects in brain glucose metabolism can predict future amyloid plaque deposition. On the other hand, early amyloid plaque deposition may predict the future occurrence of Alzheimer's disease as early as 15 years before the onset. This research project is focusing on the sequential change of the two biomarkers of brain glucose metabolism and amyloid plaque deposition and their correlation with clinical symptoms in patients with Alzheimer's disease. The subjects in this project will be including normal controls without cognitive impairment, patients with prodromal AD or AD. The relationship between functional connectivity of FDG-PET and amyloid deposition in different group of patients will be investigated. Further correlation with tau PET will be also discussed.

In the imaging process part of this project, the standard tool, SPM (Spatial Parametric Mapping) will be applied. As machine learning/deep learning methodology is gaining popularity in medical imaging research community, collaboration with artificial intelligence core laboratory at Linkou will be pursued to investigate hidden correlation between functional connectivity, amyloid plaque, progress of clinical symptoms with time that previous statistical methods may not be able to find.

ELIGIBILITY:
Inclusion Criteria:

* All the participants must meet the following criteria:

  1. Age between 55-80 years.
  2. Patients population: Diagnosed as prodromal AD or mild AD dementia based on IWG-2 criteria.
  3. Normal control population: Cognitive unimpaired individual is defined as normal control in this study. Cognitive un-impaired normal control is defined as cognitive performance in the non-impaired range for that individual, defined as not mild cognitive impairment or demented. The normal control should have their clinical dementia rating score 0 AND Cognitive Ability Screening Instrument (CASI) scores rated >50 percentile.
  4. Able to provide written informed consent with reliable caregiver in AD population. The participant should have reading ability OR 6/more years of formal education OR with working experiences.

Exclusion Criteria:

* All participants must not meet the following criteria:

  1. Already receive outpatient clinic follow-ups with diseases that may affect the cognitive evaluation or presentation that include but not limited to Parkinsonism, Parkinson's disease dementia, epilepsy, schizophrenia, major depression, major psychiatric disorders, alcohol or drug abuse, major head trauma with consciousness loss.
  2. Severe progressive or unstable systemic disease that may interfere with the follow-up and test results. These included but not limited to cancer in the past 5 years, end stage renal or liver dysfunction, clinically significant myocardial infarction (New York Heart Association Functional Classification III-IV), Active disease that received admission in the past one year and unstable angina. Other diseases that were not listed but may interfere with the follow-up or test will be judged by the principle investigator.
  3. Any treatment that suggests any of the aforementioned disease will be excluded.
  4. Depression with ongoing diagnosis and treatment, suicide idea or suicide behavior in the past 6 months.
  5. Contraindications or previously failure for receiving brain magnetic resonance imaging or PET scan.
  6. Pregnant, lactating or breastfeeding.
  7. Patients with severe liver disease (such as ALT > 3x upper limit of normal).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-03-27 (Estimated); Study Completion 2023-09-27 (Estimated)

PRIMARY OUTCOMES:
Amyloid Distribution Among Normal, Prodromal AD and AD Dementia Subjects Measured by Standardized Uptake Value Ratio (SUVR) as Assessed by 18F-AV45 amyloid PET Scan. | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital,Linkou, Taoyuan, Guishan Dist, Taiwan